CLINICAL TRIAL: NCT05095402
Title: Evaluation of the Relationship Between Lumbar Lordosis Angle and Lumbar Muscle Thickness With Non-Specific Low Back Pain
Brief Title: Biomechanics of Lumbar Region in Low Back Pain
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Ali Cihan Dagli, Principal Investigator, Karabuk University
Other Study IDs: KU-ANA-ACD-01
Record Dates: First submitted 2021-09-14; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Lumbar Lordosis Angle; Magnetic Resonance Imaging; Muscle Thickness
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to examine the relationship between non-specific low back pain (NSLBP) and lumbar lordosis angle (LLA) and lumbar muscle thickness (LMT) by evaluating magnetic resonance images (MRI) in individuals with LBP.

DETAILED DESCRIPTION:
The study included a total of 96 individuals, 43 males, and 53 females, who applied to the Department of Radiology of the Karabuk University Training and Research Hospital between March-June 2019 with complaints of LBP. Individuals' sociodemographic information and medical history were recorded using the LBP assessment form. The Oswestry LBP Disability Questionnaire was used for LBP. Thickness measurements of muscle (m.) psoas major, m. multifidus, m. quadratus lumborum and m. erector spinae were taken on MRI corresponding to the L3-L4 vertebra level. Cobb Angle method was used for LLA determination. Measurements were made in three repetitions using the Radiant DICOM viewer program, and their averages were recorded.

ELIGIBILITY:
Inclusion Criteria:

* The age range of 18-65
* Having non-specific LBP
* Volunteering to participate in the study

Exclusion Criteria:

* Having any psychiatric and mental problems
* The presence of any disc, bone, and muscular pathology in the lumbar region
* Having any previous operation on the lumbar region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included a total of 96 individuals, 43 males, and 53 females, who applied to the Department of Radiology of the Karabuk University Training and Research Hospital between March-June 2019 with complaints of LBP.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Disability caused by low back pain assessed by Oswestry Low Back Pain Disability Questionnaire | 6 months
  Low back pain disability is assessed with Oswestry Low Back Pain Disability Questionnaire.
  Oswestry Disability Index (ODI) score as a percentage is obtained from the questionnaire result.
Lumbar lordosis angle | 6 months
  * Measured with the COBB angle method as LLA degree.
  * It is determined by looking at the angle between the vertebrae forming the lumbar lordosis curvature (L1-L5).
  * All radiological measurements are performed on the RAdiant DICOM viewer program.
Muscles thickness measurements | 6 months
  * Measured on the horizontal plane corresponding to the L3-L4 level in the sagittal plane.
  * Bilaterally, the thickest parts of the muscles are measured anterior-posterior and transverse and recorded in millimetres (mm).
  * All radiological measurements are performed on the RAdiant DICOM viewer program.
  * Muscles measured are listed below:
  * m. psoas major
  * m. multifidus
  * m. erector spinae muscles
  * m. quadratus lumborum

CONTACTS AND LOCATIONS:
Overall Officials: Ali dagli, Principal Investigator — Karabuk University
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No